CLINICAL TRIAL: NCT00073866
Title: Phase I/II Trial Of Weekly Irinotecan And Docetaxel With The Addition Of Celecoxib In Advanced Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy and Celecoxib in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 01L2; NU-01L2; PHARMACIA-NU-01L2
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib
Drug: docetaxel
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may stop the growth of tumor cells by stopping blood flow to the tumor. Combining celecoxib with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of irinotecan and docetaxel when given together with celecoxib and to see how well they work in treating patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recommended phase II dose of docetaxel and irinotecan in combination with celecoxib in patients with advanced non-small cell lung cancer.
* Determine the toxic effects of this regimen in these patients.
* Determine the response rate of patients treated with this regimen.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.
* Correlate angiogenesis markers (intratumoral microvessel density and vascular endothelial growth factor [VEGF] expression and serum VEGF) and cyclooxygenase-2 expression with response and survival in patients treated with this regimen.
* Correlate UGT1A1 genotype and CYP3A4 activity with the toxic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study of docetaxel and irinotecan.

* Phase I: Patients receive docetaxel IV over 60 minutes and irinotecan IV over 30 minutes on days 1 and 8. Patients also receive oral celecoxib twice daily beginning on day 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity Cohorts of 3-6 patients receive escalating doses of docetaxel and irinotecan until the recommended phase II dose is determined. The recommended phase II dose is defined as the highest dose at which 0 of 3 or 1 of 6 patients experience dose-limiting toxicity.
* Phase II: Patients receive treatment as in phase I at the recommended phase II dose.

Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 3-70 patients (3-36 for phase I and 16-34 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer (NSCLC) meeting 1 of the following criteria:

  * Stage IV
  * Stage IIIB with a malignant pleural effusion
  * Locally recurrent and/or persistent disease after locoregional therapy with or without systemic chemotherapy
* Unidimensionally measurable disease

  * If the only site of measurable disease is in a previously irradiated area must have documented progression of disease in that area
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT less than 2.5 times upper limit of normal (ULN) (if alkaline phosphatase is normal)
* Alkaline phosphatase less than 4 times ULN (if AST and ALT are normal)

Renal

* Creatinine less than 2.0 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study treatment
* No other malignancy within the past 5 years except curatively treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No diagnosis of peptic ulcer disease or gastritis/esophagitis within the past 60 days
* No prior hypersensitivity to cyclooxygenase-2 (COX-2) inhibitors, nonsteroidal anti-inflammatory drugs (NSAIDs), salicylates, sulfonamides, or drugs formulated with polysorbate 80
* No pre-existing grade 2 or greater peripheral neuropathy
* No concurrent medical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 1 week since prior biologic therapy
* Phase I patients:

  * Any number of prior biologic therapies allowed (e.g., chimeric antibodies or kinase inhibitors)
* Phase II patients:

  * No prior biologic therapy for recurrent/metastatic disease
* No concurrent filgrastim (G-CSF)

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No prior irinotecan or docetaxel
* Phase I patients:

  * Up to 2 prior chemotherapy regimens for recurrent/metastatic disease allowed (chemonaïve patients are also eligible)
* Phase II patients:

  * At least 1 year since prior adjuvant or neoadjuvant chemotherapy for stage I-IIIA disease
  * No prior chemotherapy for recurrent/metastatic disease

Endocrine therapy

* Less than 2 weeks of cumulative oral/IV corticosteroid use within the past 3 months

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* At least 3 weeks since prior extensive-field radiotherapy for recurrent/metastatic disease

Surgery

* Recovered from prior surgery

Other

* More than 60 days since prior treatment for peptic ulcer disease or gastritis/esophagitis
* No prior NSAIDs at a frequency of more than 3 times per week for a cumulative period of more than 2 weeks within the past 30 days
* No concurrent antiepileptics, cyclosporine, aspirin, or fluconazole
* No concurrent NSAIDs
* No other concurrent COX-2 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Silver Cross Hospital, Joliet, Illinois

REFERENCES:
- [Result] Argiris A, Kut V, Luong L, Avram MJ. Phase I and pharmacokinetic study of docetaxel, irinotecan, and celecoxib in patients with advanced non-small cell lung cancer. Invest New Drugs. 2006 May;24(3):203-12. doi: 10.1007/s10637-005-3259-4. PMID 16096702